CLINICAL TRIAL: NCT07149649
Title: Magnesium Supplementation in Addition to Standard Chemo-immunotherapy in Patients With Locally Advanced Unresectable Stage III or Metastatic Stage IV Non-small Cell Lung Cancer (NSCLC). A Double-blind Randomized Multicenter Phase II/III Study.
Brief Title: Magnesium Supplementation in Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAKK 19/24
Record Dates: First submitted 2025-07-30; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Metastatic NSCLC - Non-Small Cell Lung Cancer
Keywords: Magnesium supplementation; Magnesium aspartate hydrochloride; Placebo; Non-Small Cell Lung Cancer; phase II/phase III; unresectable stage III NSCLC; metastatic stage IV NSCLC; double-blind randomized
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Aspartic Acid; levulinic acid; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo-controlled, seamless phase II/III trial. In total, 230 patients will be included in the trial - 70 patients in phase II and 160 patients in phase III.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding procedures Patient randomization into the two treatment arms is double-blind. Neither the patient nor any of the investigators who are involved in the conduct of the trial, or the analysis of the trial data have knowledge of the assigned treatment arm.
  This level of blinding is maintained throughout the conduct of the trial unless there are compelling medical or safety reasons to alleviate the unblinding.
  On the sponsor's side, the Clinical Research Associates (CRA) performing source data verification, and the CDM-DM performing data management remain blinded for the entire duration of the trial.
  Blinding is performed by the authorized pre-wholesaler upon randomization of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium (Experimental): Platinum-based chemo-immunotherapy every 3 weeks
  + Magnesium
  * intravenous at day 1 of each therapy cycle
  * peroral thrice daily (day 1-21)
  Interventions: Drug: Magnesiocard; Drug: Magnesium Diasporal
- Placebo (Active Comparator): Platinum-based chemo-immunotherapy every 3 weeks
  + Placebo
  * intravenous at day 1 of each therapy cycle
  * peroral thrice daily (day 1-21)
  Interventions: Other: Microcrystalline cellulose; Other: Isotonic saline solution 0.9%

INTERVENTIONS:
Drug: Magnesiocard — 2.5 mmol film-coated tablets in addition to standard first line therapy
  Arms: Magnesium
Drug: Magnesium Diasporal — 4 mmol IV formulation in addition to standard first line therapy
  Arms: Magnesium
Other: Microcrystalline cellulose — Placebo film-coated tablets corresponding to Magnesiocard in addition to standard first line therapy
  Arms: Placebo
Other: Isotonic saline solution 0.9% — Placebo for injection corresponding to Magnesium Diasporal in addition to standard first line therapy
  Arms: Placebo

SUMMARY:
This study investigates whether adding magnesium to the standard chemo-immunotherapy for advanced non-small cell lung cancer (NSCLC) can improve treatment outcomes. Magnesium is important for immune function, and low levels during chemotherapy are common. Participants are randomly assigned to receive either magnesium or a placebo, both as infusions and tablets. Neither the participants nor the doctors know who receives which treatment. The study compares the two groups to see if magnesium helps and how well it is tolerated.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multicenter phase II/III trial evaluates the efficacy and safety of intravenous and oral magnesium supplementation in addition to standard first-line chemo-immunotherapy in patients with unresectable stage III or metastatic stage IV non-small cell lung cancer (NSCLC).

Platinum-based chemotherapy frequently induces hypomagnesemia, which may impair T-cell mediated anti-tumor immunity and reduce the effectiveness of immune checkpoint inhibitors. This trial investigates whether correcting magnesium deficiency can enhance immune response and improve clinical outcomes.

The primary objective of the phase II portion is to assess the safety and feasibility of magnesium supplementation and its impact on PFS. If interim analysis confirms tolerability without significant additional toxicity, the trial will seamlessly expand into a phase III component with overall survival (OS) as the primary endpoint.

Secondary objectives include objective response rate (ORR), duration of response (DoR), adverse events (AEs) and serious adverse events (SAEs), health-related quality of life (HRQoL), immune-related biomarkers and magnesium levels.

Patients are randomized to receive either:

* Magnesium Arm: Standard chemo-immunotherapy + oral magnesium aspartate hydrochloride (3x/day) + intravenous magnesium sulfate on chemo days
* Placebo Arm: Standard chemo-immunotherapy + matching placebo Magnesium levels are centrally monitored via plasma and urine samples. Anti-cancer therapy follows standard of care.

  230 patients will be enrolled (70 in phase II, 160 in phase III). Eligible patients have stage IIIB/IV NSCLC, ECOG 0-1, and are scheduled for first-line chemo-immunotherapy. Key exclusions include eligibility for monotherapy, severe hypomagnesemia, or ongoing magnesium supplementation for other indications.

Statistical and Quality Considerations

The adaptive design includes an interim analysis for safety and a futility analysis for OS. Time-to-event and binary outcomes will be analyzed using standard statistical methods. Quality assurance includes eCRFs with validation checks, source data verification, SOPs, and risk-based monitoring.

Although not formally a registry, the trial employs registry-like quality control elements:

* Data validation: Real-time data entry into electronic case report forms (eCRFs) with predefined logic and range checks.
* Source Data Verification (SDV): Conducted to ensure data accuracy and completeness via comparison with medical records and source documents.
* Standard Operating Procedures: SOPs are implemented, which cover all trial operations-site initiation, data collection, patient assessments, safety reporting, and amendment handling.
* Monitoring and auditing: Central and on-site monitoring according to a risk-based monitoring plan. Sites may be audited for compliance with ICH-GCP.

This trial addresses a novel and biologically plausible mechanism of resistance to immunotherapy in NSCLC. By targeting chemotherapy-induced hypomagnesemia, the study explores a low-cost, scalable intervention with the potential to enhance immune-mediated tumor control. If successful, magnesium supplementation could represent a paradigm shift in the supportive care of patients receiving chemo-immunotherapy for advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH GCP E6 regulations before registration and prior to any trial specific procedures;
* Histologically or cytologically confirmed diagnosis of NSCLC (adeno-, squamous-, large cell carcinoma or NSCLC not otherwise specified);
* Patients planned for systemic first-line therapy with a combination of a carboplatin-based doublet chemotherapy and a PD-1 / PD-L1 targeting immune checkpoint inhibitor;
* Patients not eligible for immune checkpoint inhibitor monotherapy irrespective of PD-L1 expression;
* Locally advanced unresectable stage III or metastatic stage IV disease (defined as TNM, according to 8th edition) not eligible for curative surgery and/or definitive (curative intended) chemoradiotherapy;
* No sensitizing EGFR mutation, METex14 skipping mutation, BRAF V600E mutation, ALK/ROS1/RET, NTRK1/2 gene rearrangements, HER2 mutations, amplifications detected in primary tumor or metastases;
* Have not received prior systemic treatment for their metastatic NSCLC. Patients who received adjuvant, neoadjuvant chemotherapy or chemoradiotherapy with curative intent for nonmetastatic disease are eligible if the therapy was completed at least 12 months prior to the diagnosis of metastatic disease;
* Patients with treated and stable CNS metastases are eligible, provided they meet the following criteria:

  * No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
  * No stereotactic radiation or whole-brain radiation within 14 days prior to registration.
* Patients with known HIV-infection, who are at low risk of AIDS-related outcomes, are eligible, provided they meet the following criteria:

  * CD4+ T-cell counts are ≥ 350 cells/ųL
  * No history of AIDS-defining opportunistic infection within past 12 months
  * Patients have been on antiretroviral therapy (ART) for > 4 weeks before registration and have a HIV viral load < 400 copies/mL;
* Patients with a prior malignancy and treated with curative intention are eligible if the treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence;
* Measurable disease per RECIST v1.134);
* Age ≥ 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* Adequate bone marrow function as per local guidelines;
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST and ALT ≤ 2.5 x ULN, or ≤ 5 x ULN under the assumption that abnormal values are a result of NSCLC;
* Adequate renal function defined by stable estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m2 (according to CKD-EPI formula);
* Women of childbearing potential must use highly effective contraception (see chapter 9.4), are not pregnant or lactating and agree not to become pregnant during trial treatment and until 6 months after the last dose of investigational drug. A negative pregnancy test before inclusion into the trial is required for all women of childbearing potential.
* Men agree not to donate sperm or to father a child during trial treatment and until 6 months after the last dose of investigational drug.

Exclusion Criteria:

* Plasma magnesium concentration < 0.4 mmol/l or > 1.2 mmol/L
* Treatment with any anti-cancer therapy within 21 days prior to registration (excluding hormonal therapy or anti-cancer surgery). Any previous anti-cancer therapy must have been administered with curative intent;
* Treatment with radiotherapy within 14 days prior to registration (except for local pain control);
* Patients planned for cisplatin-based chemo-immunotherapy;
* Treatment with any other experimental drug within 28 days of registration;
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia);
* Atrioventricular (AV) block of any degree unless being treated with cardiac pacemakers;
* Bradycardia <40/min at steady state;
* Active chronic Hepatitis C or Hepatitis B infection or any uncontrolled active systemic infection, needing antibiotic treatment within 14 days before registration;
* Known history of tuberculosis, known history of relevant primary immunodeficiency, known history of allogeneic organ transplant, receipt of live attenuated vaccine within 28 days prior to registration;
* Diagnosis of myasthenia gravis;
* Concomitant or prior use of immunosuppressive medication within 28 days before registration, with the exceptions of:

  * intranasal and inhaled corticosteroids
  * systemic corticosteroids ≤ 10 mg/day of prednisone, or a dose equivalent corticosteroid,
  * premedication for chemotherapy;
* Prior treatment with peroral or intravenous magnesium 14 days prior to registration;
* Patient not willing to stop the use of peroral magnesium treatment including over the counter or lifestyle products;
* Any concomitant drugs contraindicated for use with the trial drug according to the approved product information;
* Known hypersensitivity to any of the trial drugs;
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2035-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint of Phase II part: Progression-free survival (PFS) | From randomization to PD or death, up to 10 years
  PFS defined as time from randomization to progression according to RECIST 1.1 criteria or death. Patients not experiencing an event will be censored at the date of the last available assessment before initiation of a new anti-cancer treatment, if any.
Primary endpoint of Phase III part: Overall survival (OS) | From randomization to PD or death, up to 10 years
  OS defined as the time from randomization until death due to any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.

SECONDARY OUTCOMES:
Toxicity - Intermediate endpoint for the adaptive decision to expand, or not, into a Phase III | All adverse events: from baseline until end of treatment, deaths: until end of follow-up, up to 10 years
  Immune related adverse events (irAEs) ≥ Grade 3 according to NCI CTCAE v5.0
Number of participants discontinued any treatment component. | from baseline until end of treatment, deaths: until end of follow-up, up to 10 years
  Tolerability - Intermediate endpoint for the adaptive decision to expand, or not, into a Phase III. Discontinuation of any treatment component (chemotherapy and/or immunotherapy) within the first 4 cycles of treatment
Event-free survival (EFS) | From randomization to PD, 2nd tumor or death, up to 10 years
  EFS is defined as time from registration to one of the following events, whichever occurs first:
  * Relapse or progression according to RECIST 1.1 criteria
  * Second tumor
  * Death due to any cause Patients not experiencing an event will be censored at the date of the last available assessment before initiation of a new anti-cancer treatment, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Lötscher, MD, PhD, Study Chair — CH - Universitätsspital Basel; Sacha Rothschild, Prof MD, PhD, Study Director — CH - Kantonsspital Baden; Christoph Hess, Prof MD, PhD, Study Director — CH - Universitätsspital Basel
Locations (11):
- Switzerland (11):
  - Tumorzentrum Aarau - Hirslanden TZA, Aarau
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - St. Claraspital, Basel
  - Universitätsspital Basel, Basel
  - Kantonsspital Graubuenden, Chur
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Winterthur